CLINICAL TRIAL: NCT05863572
Title: Strengthening Care in Collaboration With People With Lived Experience of Psychosis in Uganda
Acronym: SCAPE-U
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: YouBelong Uganda (Unknown); Butabika National Referral Hospital (Unknown)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS2327ES
Record Dates: First submitted 2023-04-12; First posted 2023-05-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — House Calls

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are masked to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Training primary care workers in diagnosis and treatment; training community health workers in detection and referral.
  Interventions: Other: Primary care health worker training; Other: Community Health Workers Training
- Strengthening care in collaboration with people with lived experience of psychosis in Uganda (Experimental): Trainings done in collaboration with people with lived experience of psychosis; as well as additional home visits conducted by people with lived experience of psychosis.
  Interventions: Other: Primary care health worker training; Other: Community Health Workers Training; Other: Home visits

INTERVENTIONS:
Other: Primary care health worker training — Training primary care workers to detect and treat psychosis.
Other: Community Health Workers Training — training community health workers in detection and referral
Other: Home visits — home visits conducted by people with lived experience of psychosis
  Arms: Strengthening care in collaboration with people with lived experience of psychosis in Uganda

SUMMARY:
Background: Mental health services are most effective and equitable when designed, delivered, and evaluated in collaboration with people with lived experience of mental health conditions. Unfortunately, people with lived experience are rarely involved in health systems strengthening or are limited to specific components (e.g., peer helpers) rather than multi-tiered collaboration in the continuum of health services (e.g., ranging from home- to community- to clinic-based services). Moreover, programs that do involve people with lived experience, typically involve people with a history of a substance use conditions or common mental disorders. In contrast, the collaboration of people with lived experience of psychosis is especially rare. A pilot cluster randomized controlled trial will be conducted in urban and peri-urban areas around Kampala, Uganda, to evaluate the benefits of an implementation strategy for mental health services with engagement of people with lived experience of psychosis throughout the home-to-community-to-clinic care continuum, this is a hybrid type-III implementation-effectiveness pilot focusing on the differences in implementation strategy. This implementation strategy, entitled "Strengthening CAre in collaboration with People with lived Experience of psychosis in Uganda", will include training people with lived experience of psychosis using PhotoVoice and other methods to participate at three levels: in-home services, community engagement, and primary health care facilities. The investigators will compare a standard task-sharing implementation arm using training by mental health specialists with an experimental implementation arm that includes collaboration with people with lived experience. The primary objective is to evaluate the feasibility and acceptability of this strategy in the context of assuring safety and wellbeing of people with lived experience of psychosis who collaborate in health systems strengthening. By collaborating on health systems strengthening across these multiple levels, we foresee a more in-depth contribution that can lead to rethinking how best to design and deliver care for people with lived experience of psychosis. Successful completion of this pilot will be the foundation for a fully powered trial to evaluate the benefits of multi-level collaboration with people with lived experience of psychosis.

DETAILED DESCRIPTION:
The aim of the current study is to conduct a pilot cluster randomized controlled trial to determine feasibility and acceptability of people with lived experience of psychosis collaborating in training primary care and community health care workers and co-delivering services in the home. This pilot study will consist of two trial arms: - Training- As- Usual vs the experimental arm. It will be implemented across three-tiers - in primary health care, community, and home settings. The pilot will also determine the parameters needed for appropriate design and implementation of a fully-power future cluster randomized controlled trial.

Objective 1 - To assess the feasibility and acceptability of the implementation strategy from the perspective of people with lived experience of psychosis, family members and primary and community care providers.

Objective 2 - To demonstrate proof-of-concept for the benefit of the implementation strategy for service users (i.e., patients with psychosis receiving primary care services) and their families, including changes in psychosis symptoms, quality of life, frequency of hospitalization and the potential impacts on family members.

Objective 3 - To evaluate changes in health systems outcomes in terms of primary care provider knowledge, attitudes, competency in psychosis diagnosis and management, accuracy of diagnosis and fidelity to treatment guidelines in actual care settings as well as trial procedures.

Objective 4: To evaluate costing, recruitment and retention, and data collection procedures and protocols to determine the optimal design for a future fully powered cluster Randomized Controlled Trial.

Objective 5: To establish and demonstrate ethics and safety in collaborating with service users.

ELIGIBILITY:
Inclusion Criteria:

1. Facilitators of the implementation strategy:

   1. At least 18 years of age
   2. Confirmed diagnosis of a primary psychotic disorder (e.g., schizophrenia) by a psychiatrist or psychiatric clinical officer
   3. Completion of the YouBelongHOME (YBH) program
   4. Provision of informed consent,
   5. Fluency in the local language (Luganda)
   6. Good functioning with respect to performance of daily chores,engagement with family members, comprehension and community participation as assessed by the YBH team
   7. A supportive family member.
2. Primary care providers:

   1. Provides primary care in health facility of Kampala/Wakiso District
   2. Selected by facility in-charge
3. Community health workers

   1. Provides community based health service in health facility where primary care providers are trained (from Kampala/Wakiso district)
   2. Selected by facility in-charge
4. Patients (Primary beneficiaries)

   1. Persons diagnosed with psychosis at a primary health care facility in Kampala/Wakiso District; For this study, a diagnosis of psychosis will include the following diagnoses according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5):schizophrenia spectrum and other psychotic disorders [brief psychotic disorder, schizophreniform disorder, schizoaffective disorder, schizophrenia, and organic psychosis (i.e., psychosis secondary to a medical condition such as HIV or an alcohol- or substance-use disorder)];bipolar affective disorder and related disorders;
   2. Ability of the patient or responsible surrogate to consent to study enrolment and procedures;
   3. Persons eligible for outpatient management of psychosis
5. Family members a. Family member or caregiver of the patients above.

Exclusion Criteria:

1. Facilitators of the implementation strategy:

   a. Inability to provide informed consent.
2. Primary care providers:

   None
3. Community health workers:

   None
4. Patients

   1. Persons diagnosed with psychosis requiring inpatient management/services; and
   2. Persons for whom consent for participation in the study cannot be obtained.
   3. Patients found to be severely ill beyond the capacity of the health facility to treat.
5. Family members a. Family members who doesn't provide consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Symptoms of Schizophrenia (PANSS) scale | baseline - immediately after enrollment
  Symptoms of Psychosis, minimum = 0, maximum = 56, higher score is worse
Positive and Negative Symptoms of Schizophrenia (PANSS) scale | 4 months post enrollment
  Symptoms of Psychosis, minimum = 0, maximum = 56, higher score is worse
Positive and Negative Symptoms of Schizophrenia (PANSS) scale | 8 months post enrollment
  Symptoms of Psychosis, minimum = 0, maximum = 56, higher score is worse

SECONDARY OUTCOMES:
World Health Organization Quality of Life-Brief Scale | immediately after enrollment
  Brief quality of life scale, minimum = 0, maximum = 100, Higher score refers to better quality of life
World Health Organization Quality of Life-Brief Scale | 4 months post enrollment
  Brief quality of life scale, minimum = 0, maximum = 100, Higher score refers to better quality of life
World Health Organization Quality of Life-Brief Scale | 8 months post enrollment
  Brief quality of life scale, minimum = 0, maximum = 100, Higher score refers to better quality of life
Service user collaboration checklist | immediately after enrollment
  Benefits and challenges of service users' collaboration, minimum = 12, maximum = 48, higher number refers to strong collaboration experience
Service user collaboration checklist | 4 months post enrollment
  Benefits and challenges of service users' collaboration, minimum = 12, maximum = 48, higher number refers to strong collaboration experience
Service user collaboration checklist | 8 months post enrollment
  Benefits and challenges of service users' collaboration, minimum = 12, maximum = 48, higher number refers to strong collaboration experience
EuroQuality of Life 5-Dimension 5-Level | immediately after enrollment
  Quality of Life (for health economics analyses), minimum = 5, maximum=25, higher score is worse
EuroQuality of Life 5-Dimension 5-Level | 4 months post enrollment
  Quality of Life (for health economics analyses), minimum = 5, maximum=25, higher score is worse
EuroQuality of Life 5-Dimension 5-Level | 8 months post enrollment
  Quality of Life (for health economics analyses), minimum = 5, maximum=25, higher score is worse
Discrimination and Stigma Scale-Brief version | immediately after enrollment
  Stigma experienced by persons living with mental illness, minimum = 0, maximum = 33, Higher score refers to higher experience of stigma
Discrimination and Stigma Scale-Brief version | 4 months post enrollment
  Stigma experienced by persons living with mental illness, minimum = 0, maximum = 33, Higher score refers to higher experience of stigma
Discrimination and Stigma Scale-Brief version | 8 months post enrollment
  Stigma experienced by persons living with mental illness, minimum = 0, maximum = 33, Higher score refers to higher experience of stigma
Social Inclusion Scale | immediately after enrollment
  Social Inclusion of service users, minimum = 10, maximum = 50, Higher score refers to better experience of social inclusion
Social Inclusion Scale | 4 months post enrollment
  Social Inclusion of service users, minimum = 10, maximum = 50, Higher score refers to better experience of social inclusion
Social Inclusion Scale | 8 months post enrollment
  Social Inclusion of service users, minimum = 10, maximum = 50, Higher score refers to better experience of social inclusion
Hospitalization Record | immediately after enrollment
  no minimum or maximum, score is total number of days patient was hospitalized during study period
Hospitalization Record | 4 months post-enrollment
  no minimum or maximum, score is total number of days patient was hospitalized during study period
Hospitalization Record | 8 months post enrollment
  no minimum or maximum, score is total number of days patient was hospitalized during study period
Client Service Receipt Inventory | immediately after enrollment
  Costs of care to patients, there is no maximum or minimum score, the outcome is total cost for patient to get healthcare
Client Service Receipt Inventory | 4 months post enrollment
  Costs of care to patients, there is no maximum or minimum score, the outcome is total cost for patient to get healthcare
Client Service Receipt Inventory | 8 months post enrollment
  Costs of care to patients, there is no maximum or minimum score, the outcome is total cost for patient to get healthcare
Family Interview Schedule-Impact on Caregivers | immediately after enrollment
  Impact on family members and caregivers of people with mental illness, minimum = 0, maximum = 48, higher score means higher burden on the families
Family Interview Schedule-Impact on Caregivers | 4 months post enrollment
  Impact on family members and caregivers of people with mental illness, minimum = 0, maximum = 48, higher score means higher burden on the families
Family Interview Schedule-Impact on Caregivers | 8 months post enrollment
  Impact on family members and caregivers of people with mental illness, minimum = 0, maximum = 48, higher score means higher burden on the families
Community Health Workers: Social Distance Scale | pre training
  Attitudes of community health workers towards people with psychosis, 12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Community Health Workers: Social Distance Scale | immediately after training
  Attitudes of community health workers towards people with psychosis, 12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Community Health Workers: Assessment tool | monthly throughout the study period : average of 8 months, However accuracy check during SCID diagnosis check
  Accuracy of detection, no score - will check if their detection matches with the gold standard - Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders 5
Community Health Workers: Village health team referral | monthly throughout the study period (average of 8 months), starts immediately after training
  no maximum or minimum, outcome is the number of patients referred by community health workers to the health post
Community Health Workers: Village health team referral with psychosis | monthly throughout the study period (average of 8 months), starts immediately after training
  no maximum or minimum, outcome is the number of patients diagnosed with psychosis by PCP and referred by community health workers to the health post
Primary care workers: Social Distance Scale | pre training
  12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Primary care workers: Social Distance Scale | immediately after training
  12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Primary care workers: Social Distance Scale | final supervision: 8 months post training
  12-item scale of willingness to interact with persons with mental illness, minimum = 0, maximum = 72, higher score is worse outcome
Primary care workers: Mental health Gap Action Program Knowledge | pre training
  Multiple-choice assessment from mental health Gap Action Programme training materials; minimum = 0, maximum = 100, higher is better outcome
Primary care workers: Mental health Gap Action Program Knowledge | immediately after training
  Multiple-choice assessment from mental health Gap Action Programme training materials; minimum = 0, maximum = 100, higher is better outcome
Primary care workers: Mental health Gap Action Program Knowledge | final supervision: 8 months post training
  Multiple-choice assessment from mental health Gap Action Programme training materials; minimum = 0, maximum = 100, higher is better outcome
Primary care workers: Enhancing Assessment of Common Therapeutic factors for Psychosis | pre training
  Observed structured clinical evaluation using a standardized role play, minimum score = 0, maximum = 100, higher scores are better
Primary care workers: Enhancing Assessment of Common Therapeutic factors for Psychosis | immediately after training
  Observed structured clinical evaluation using a standardized role play, minimum score = 0, maximum = 100, higher scores are better
Primary care workers: Enhancing Assessment of Common Therapeutic factors for Psychosis | final supervision - 8 months post training
  Observed structured clinical evaluation using a standardized role play, minimum score = 0, maximum = 100, higher scores are better
Health Facility Record | pre training
  no minimum or maximum, score is the total number of patient diagnosed with psychosis : clinical records reviewed by Research Assistants
Health Facility Record | immediately after training
  no minimum or maximum, score is the total number of patient diagnosed with psychosis : clinical records reviewed by Research Assistants
Health Facility Record | final supervision - 8 months post training
  no minimum or maximum, score is the total number of patient diagnosed with psychosis : clinical records reviewed by Research Assistants
Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders 5 | 3 months post patient enrollment
  Accuracy of patient diagnosis by study mental health specialist

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Kohrt, MD, PhD, Principal Investigator — George Washington University; Byamah Mutamba, MD, PhD, Principal Investigator — YouBelong Uganda
Locations (1):
- YouBelong Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. No plan for feasibility study.

REFERENCES:
- [Derived] Mutamba BB, Rai S, Semakula L, Cappo D, Asher L, Gwaikolo W, Kohrt BA. Strengthening care in collaboration with people with lived experience of psychosis in Uganda (SCAPE-U): A protocol for a cluster randomized controlled feasibility trial. Pilot Feasibility Stud. 2025 Jul 21;11(1):103. doi: 10.1186/s40814-025-01684-8. PMID 40691846